CLINICAL TRIAL: NCT03250897
Title: Phenotypic Characterization of Alveolar Macrophages 2016
Brief Title: Phenotypic Characterization of Alveolar Macrophages 2016 (Caract-Aires-2016)
Acronym: Caract-Aires
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_3055_Caract-Aires-2016
Record Dates: First submitted 2017-08-11; First posted 2017-08-16 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Lung Diseases
Keywords: Alveolar macrophages; Blood monocyte-derived macrophages; FACS analysis; Broncho-alveolar lavage fluids; Non-infectious lung diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Broncho-alveolar lavage fluids of patients with non-infectious lung diseases
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to investigate by flow cytometry the phenotype of alveolar macrophages (AMs) isolated from patients with non-infectious lung diseases.

DETAILED DESCRIPTION:
Although alveolar macrophages (AMs) represent the main immune cell population in the human lungs, consensus on their phenotypic characterization is still missing.

Current translational protocols use human AMs obtained by invasive methods (broncho-alveolar lavage and lung biopsy) or differentiate macrophages from blood monocytes cultured in the presence of growth factors such as macrophage colony-stimulating factor (M-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF). The group has already published the phenotypic and functional comparison of human blood monocyte-derived macrophages differentiated with M-CSF or GM-CSF. Aim of this study is to use a multi-staining flow cytometry (FACS analysis) to better characterize the phenotype of AMs isolated from broncho-alveolar lavage fluids of patients affected by non-infectious lung diseases. The FACS profiles of AMs will be further compared to the phenotypic profile of blood monocyte-derived macrophages differentiated in the presence of GM-CSF or M-CSF. The results of this study will allow to define the most valid in vitro model of AMs in a non-infectious setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by non-infectious lung diseases and for whom a broncho-alveolar lavage is scheduled for their medical care in the pulmonary division
* Patient Information leaflet provided
* Written informed consent of the patient

Exclusion Criteria:

* A suspected respiratory infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by non-infectious lung diseases older than 18 years
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
To investigate by flow cytometry the phenotype of alveolar macrophages (AMs) isolated from broncho-alveolar lavage fluids of patients with non-infectious lung diseases. | 1 year
  Characterization of membrane proteins by multi-staining flow cytometry (FACS analysis)

SECONDARY OUTCOMES:
To compare the phenotypic profile of AMs from broncho-alveolar lavage fluids of patients with non-infectious lung diseases to that of blood monocyte-derived macrophages differentiated in the presence of GM-CSF or M-CSF and obtained from healthy donors | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Jouneau, Professor, Principal Investigator — Rennes University Hospital
Locations (1):
- Pneumology Division, Rennes, France